CLINICAL TRIAL: NCT00002227
Title: A Phase II, Open-Label, Multicenter Study to Characterize the Effectiveness and Safety of Efavirenz in Combination With Stavudine and Lamivudine in Antiretroviral Therapy-Naive HIV-Infected Patients
Brief Title: A Study of Efavirenz in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dupont Merck (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 281C; DMP 266-043
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; Lamivudine; Reverse Transcriptase Inhibitors; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Efavirenz
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give efavirenz plus stavudine plus lamivudine to patients who have never taken anti-HIV drugs.

DETAILED DESCRIPTION:
Patients will be given combination treatment with efavirenz, stavudine, and lamivudine.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented diagnosis of HIV infection with plasma HIV-RNA greater than or equal to 10,000 copies/ml.
* Life expectancy of at least 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current bilateral peripheral neuropathy greater than or equal to Grade 2.
* Proven or suspected acute hepatitis due to any cause.
* Recurrent episodes of moderate to severe diarrhea, or vomiting lasting for more than 4 days within 3 months prior to dosing.
* Hypersensitivity to any component of the formulation of efavirenz, stavudine, or lamivudine.
* Any clinically significant laboratory findings obtained during the screening evaluation (see laboratory values).
* Any clinically significant disease (other than HIV infection) or clinically significant findings found during the screening of medical history or physical examination.
* Any malignancy that requires systemic therapy.
* Any active AIDS-defining opportunistic infection or disease.

Concurrent Medication:

Excluded:

Astemizole, cisapride, clarithromycin, ketoconazole, itraconazole, midazolam, rifabutin, rifampin, terfenadine, thalidomide, triazolam, vincristine, zalcitabine or any medications contraindicated for concomitant use with stavudine or lamivudine as described in the current information package insert.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* A life expectancy of less than 12 months.
* Difficulty swallowing capsules/tablets.
* Inability to communicate effectively with study personnel.

Prior Medication:

Excluded:

* Any other experimental drug within 30 days of introducing study treatment.
* Vaccination within 3 weeks of screening visit.
* Any prior antiretroviral therapy.
* Interferon started within 30 days of initiating study treatment.

Risk Behavior:

Excluded:

Current alcohol or illicit drug use which interferes with patient's ability to follow study regimen.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Richard Elion, Washington D.C., District of Columbia
  - The Whitman Walker Clinic, Washington D.C., District of Columbia
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Remington Davis Inc, Columbus, Ohio
  - The Milton S Hersey Med Ctr / Div of Hematology, Hershey, Pennsylvania
  - Coastal Carolina Research Ctr, Mt. Pleasant, South Carolina
  - Montrose Clinic, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia